CLINICAL TRIAL: NCT05336032
Title: Ethnic Variability in Glycemic and Hunger Satiety Response to Rice in Overweight Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Dr.Amena Sadiya, Manager Dietetics, Rashid Centre for Diabetes and Research
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: SKMCA
Record Dates: First submitted 2022-03-25; First posted 2022-04-20 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Glycemic Response
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral glucose tolerance test (Active Comparator): The volunteer will be performing the standardized oral glucose tolerance test with 75 gm of glucose. After an overnight fast of 10 hours the venous blood will be collected at fasting, 30, 60 and 120 minutes post-prandial and hunger-satiety scale recorded at the same interval.
  Interventions: Other: Food (rice)
- Post prandial response to Rice (Experimental): The participants will be served cooked basmati rice (70-gram available glucose). After an overnight fast of 10 hours the venous blood will be collected at fasting, 30, 60 and 120 minutes post-prandial and hunger-satiety scale recorded at the same interval.
  Interventions: Other: Food (rice)

INTERVENTIONS:
Other: Food (rice) — Cooked rice with 75 gm carbohydrate

SUMMARY:
Evidence has./ indicated increased risk of type 2 diabetes with white rice consumption in Asian population. It is shown that glycemic response to carbohydrate-containing food may differ in people of different ethnicities. The large increment in glucose concentration induced by high glycemic index food often exaggerates the body's anabolic responses, which facilitates the overproduction of insulin and eventually results in pancreatic beta-cell failure, causing type 2 diabetes mellitus.

Given that rice is the staple food of Asians and Emiratis, and extent to which rice influences postprandial glycemia could have potential relevance in the prevention and treatment of diabetes.

In this study, the investigators intend to compare the glycemic and hunger satiety response to rice among overweight Emiratis, Asians, and Caucasian. The primary objective of the study is to compare the glycemic (glucose) and hunger satiety (hormone ghrelin and peptide YY) response to glucose and rice among overweight Emiratis, Asians, and Caucasians.

DETAILED DESCRIPTION:
An increased incidence of type 2 diabetes is a characteristic feature of populations that have undergone nutritional transition. First seen in the developed Western world, the same pattern is now being observed in Middle East and Asian countries, and United Arab Emirates (UAE) is one of them. Although overconsumption of energy and accumulation of excess body fat is a common cause of type 2 diabetes, diet almost certainly has other unknown effects, and specific foods with particular adverse effects may have a direct role in the development of type 2 diabetes. Recent meta-analysis and systematic reviews have indicated increased risk of type 2 diabetes with white rice consumption in Asian population. It is shown that glycemic response to carbohydrate-containing food may differ in people of different ethnicities. Previous studies have shown that identical carbohydrate loads elicit 2-3 times larger postprandial peaks in Asians compared to Caucasians. Although there are comparative studies reported in this region. The large increment in glucose concentration induced by high glycemic index food often exaggerates the body's anabolic responses, which facilitates the overproduction of insulin and eventually results in pancreatic beta-cell failure, causing type 2 diabetes mellitus.

Given that rice is the staple food of Asians and Emiratis, and extent to which rice influences postprandial glycemia could have potential relevance in the prevention and treatment of diabetes.

In this study, the investigators intend to compare the glycemic and hunger satiety response to rice among overweight Emiratis, Indian, and Caucasian.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to comply with study procedures and given written consent

  * Asian/Emirati/European ethnicity (both parents same ethnicity)
  * Body mass index between 24.9-29.9 kg/m2
  * Age 18-55 years
  * Fasting blood glucose <6.0 mmol/L

Exclusion Criteria:

* • Subjects with chronic diseases, including diabetes, untreated hypertension, renal impairment, gastrointestinal problems, post bariatric, known eating disorders

  * Use of medication affecting glucose metabolism
  * Recent changes in weight of > 5 % ove the past 3 months
  * On antibiotics for the past 3 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
To compare the post prandial glucose response to oral glucose and rice among Emiratis, Asians, and Caucasian overweight adults | 2 hours
  post prandial glucose response at baseline, 30, 60, 120 minutes, oral glucose tolerance test (75 gm glucose) Vs. post prandial glucose response to rice test (75 gm available glucose)
To compare the post prandial insulin response to oral glucose and rice among Emiratis, Asians, and Caucasian overweight adults | 2 hours
  post prandial insulin response at baseline, 30, 60, 120 minutes, oral glucose tolerance test (75 gm glucose) Vs. post prandial insulin response to rice test (75 gm available glucose)

SECONDARY OUTCOMES:
To compare the post prandial hunger (ghrelin hormone) to oral glucose and rice among Asian, Emirati and European Caucasian overweight adults | 2 hours
  post prandial ghrelin hormone response at baseline, 30, 60, 120 minutes, with oral glucose tolerance test (75 gm glucose) Vs. post prandial ghrelin hormone response to rice test (75 gm available glucose)
To compare the post prandial satiety (peptide-yy hormone) to oral glucose and rice among Asian, Emirati and European Caucasian overweight adults | 2 hours
  post prandial peptide -yy hormone response at baseline, 30, 60, 120 minutes, with oral glucose tolerance test (75 gm glucose) Vs. post prandial peptide-yy hormone response to rice test (75 gm available glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Rashid Centre for Diabetes and Research, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided